CLINICAL TRIAL: NCT06160193
Title: A Randomized Controlled Multicenter Trial on the Effectiveness and Acceptability of a Brief Behavioral Training for Parents of Children With Behavioral Difficulties in Primary Care Settings
Brief Title: Brief Parent Training for Children With Behavioral Difficulties in Primary Care Settings
Acronym: PAINT-POH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Accare (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METc 2023/359; PPO-RF-32 (Other Grant/Funding Number: PPO Researchfonds)
Record Dates: First submitted 2023-11-29; First posted 2023-12-07 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-01

CONDITIONS: Behavioral Difficulties
Keywords: Parent Training; Behavioral Parent Training; Brief Parent Training; Individually-Tailored; Behavioral Difficulties; Disruptive Behavior; Behavior Problems; Children; Randomized Controlled Trial; Brief Treatment; Primary Care Setting; Primary Care; General Practitioners' Practices; Behavioral Problems; Problem Behaviors
MeSH Terms: conditions — Problem Behavior; Mental Disorders

STUDY DESIGN:
Intervention Model Description: We will conduct a two-armed randomized controlled trial. Children and their parents will be randomly assigned (simple and parallel randomization) to (a) the intervention condition in which parents receive the brief parent training and may receive care as usual, or (b) the control condition in which parents may receive care as usual only.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief behavioral parent training with optional care as usual (Experimental): A brief, individualized, three-session parent training that exists of two (bi)weekly individually tailored training sessions of 120 minutes, and a third session of 60 minutes. Parents and children may receive care as usual as well. Care as usual may include all mental health care that is usually provided within or outside (e.g., at a child mental healthcare institution or at school) the general practitioners practice, except from pharmacological treatment for children's behavioral difficulties and/or behavioral parent training/support, up until the first posttreatment assessment (T1). Care as usual can also imply that there is no support or treatment.
  Interventions: Behavioral: Brief behavioral parent training with optional care as usual; Other: Care as usual
- Care as usual only (Active Comparator): Care as usual may include all mental health care that is usually provided within or outside (e.g., at a child mental healthcare institution or at school) the general practitioners practice, except from pharmacological treatment for children's behavioral difficulties and/or behavioral parent training/support, up until the first posttreatment assessment (T1). Care as usual can also imply that there is no support or treatment.
  Interventions: Other: Care as usual

INTERVENTIONS:
Behavioral: Brief behavioral parent training with optional care as usual — A brief behavioral parent training program that combines individually-tailored stimulus control and contingency management techniques to treat children's behavioral difficulties in two (bi)weekly training sessions of 120 minutes, and a third session of 60 minutes, in which the training will be evaluated and maintenance training will be provided.
  Other Names: The PAINT-P program; Brief parent training
  Arms: Brief behavioral parent training with optional care as usual
Other: Care as usual — Care as usual may include all mental health care that is usually provided within or outside (e.g., at a child mental healthcare institution or at school) the general practitioners practice, except from pharmacological treatment for children's behavioral difficulties and/or behavioral parent training/support, up until the first posttreatment assessment (T1). Care as usual can also imply that there is no support or treatment.
  Other Names: CAU

SUMMARY:
The goal of this two-armed randomized controlled trial is to investigate the effectiveness of a new, individually tailored, brief behavioral training for parents of children with behavioral difficulties in general practitioners' practices.

The main questions the study aims to examine are:

1. The short-term effectiveness of a brief and individually-tailored, behavioral parent training program in primary care settings on the severity of four daily rated target behaviors in specific home situations, compared to care as usual (CAU).
2. The short-term effectiveness of the brief parent training compared to CAU on secondary outcome measures: severity of the same four daily rated target behaviors in other home situations, severity of child disruptive behaviors, number of child disruptive behaviors perceived as troublesome by the parents, overall impairment of child behavioral difficulties, impact of child behavioral difficulties on the relationship with parents, parenting behaviors, parenting stress and parenting self-efficacy.
3. The longer-term outcomes (three month follow-up) of the brief parent training program on primary and secondary outcomes.
4. The satisfaction and acceptability of the brief parent training program in primary care settings as perceived by parents and child mental health workers.

Parents will be randomly assigned (simple and parallel randomization) to (a) the intervention condition in which parents receive three sessions of brief parent training and may receive CAU, or (b) the control condition in which parents may receive CAU. The brief parent training provides parents with individually tailored stimulus control and contingency management techniques to treat children's behavioral difficulties in two (bi)weekly training sessions of two hours and a third session of one hour in which the training will be evaluated and maintenance training will be provided. CAU may include any support or treatment as regularly provided by general practices, mental health care centers, schools and/or other organizations, except from pharmacological treatment for children's behavioral difficulties and/or behavioral parent training/support. CAU may also imply that there is no support or treatment. After the first posttreatment assessment (T1) parents in the control condition will be offered the brief parent training as well.

DETAILED DESCRIPTION:
STUDY DESIGN

We will conduct a two-armed randomized controlled trial. Children and their parents will be randomly assigned (simple and parallel randomization) to (a) the intervention condition in which parents receive the brief parent training and may receive care as usual, or (b) the control condition in which parents may receive care as usual only.

The trial will take place in several general practitioners' practices throughout the Netherlands. The brief parent training will be provided by child mental health workers (in Dutch: praktijkondersteuners GGZ kind en jeugd).

TIME FRAME

December 2023: start recruitment, screening and inclusion of parents and children, start running interventions.

December 2023 until September 2025: ongoing contacts with general practitioners practices; recruitment, screening, and inclusion of children; run interventions and conduct measurements; supervision of therapists; fidelity checks; other project management activities.

September 2025 until September 2027: data-analysis, dissemination of results, implementation activities.

SAMPLE SIZE ASSESSMENT

In our prior study conducted in specialized mental health care with experienced behavioral therapists (all with MA degree), we found moderate short-term effects on momentary assessed (i.e., daily) ratings of behavioral difficulties compared to waitlist (range of Cohen's d .54 to .66; Hornstra et al., 2021). The current trial will take place in a less specialized setting, with a more heterogenous group of mental health care providers (also BA degree), who are generally less educated in behavioral therapy. Therefore, we expect the effect to be between small to moderate (d = 0.35).

A power analysis has been performed using G*Power software (Faul, 2007). Based on an effect size of d = 0.35, two groups and two repeated measures (T0 and T1 for short term effectiveness, with r = .60 between-measurement correlation), a power of .80 and alpha = 0.05, we would need 27 participants per group, resulting in a total of 54 participants. Given that our data is clustered, we multiplied our total sample with 110%, resulting in a total number 60 participants (Twisk et al., 2013).

TREATMENT OF SUBJECTS - BRIEF PARENT TRAINING PROGRAM (INTERVENTION CONDITION)

The brief parent training program consists of three sessions. The first two sessions will take 120 minutes and the third session will take 60 minutes. All three sessions will be spread over a maximum of six weeks. In between sessions, parents are asked to read some materials and implement the plan as created during the session at home.

The brief parent training program uses the behavioral techniques that were identified as effective for behavioral difficulties in a microtrial of our group (Hornstra et al., 2021) and the broader literature (Kaminski et al., 2008; Leijten et al., 2019; Leijten et al., 2021). The program combines the stimulus control and contingency management techniques that, separately, reduced behavioral difficulties in the microtrial.

In the screening phase, parents indicate which four, daily occurring, target behaviors they prefer to address in the training. They also indicate in which specific situations these behaviors mostly occur. The selected behaviors and situations will be sent to the child mental health worker. Out of the four target behaviors, two will be addressed during the training.

The first session consists of four steps. First, psycho-education will be provided on executive function problems and motivational issues that may occur in children with behavioral difficulties. Second, using functional analyses, the child mental health worker and parents will determine which of the available techniques may address the first target behavior in the specific situation. Third, the child mental health worker and parents make an action plan for the target behavior in the specific situation, in which these techniques are included and explained to the parents. Fourth, the action plan will be practiced using role play and the parents are instructed to implement the action plan as soon as possible at home. In the second session, the plan that was made in the previous session will first be evaluated. Thereafter, the same steps will be repeated for a second problem behavior. In the third session, the child mental health worker and parents will evaluate both plans and discuss how to maintain and generalize the behavioral techniques that proved to work.

Parents allocated to the intervention condition may receive care as usual as well.

TREATMENT OF SUBJECTS - CARE AS USUAL (CONTROL CONDITION)

Care as usual may include all mental health care that is usually provided within or outside (e.g., at a child mental healthcare institution or at school) the general practitioners' practice, except from pharmacological treatment for children's behavioral difficulties and/or behavioral parent training/support, up until the first posttreatment assessment (T1). Care as usual can also imply that there is no support or treatment.

METHODS

Demographic information about the child and parents will be collected with a self-composed questionnaire, with questions about the age and gender of the child, household composition, native country of the child and parents, school type of the child, educational background of the parents, (possible) mental disorders of the child, and mental healthcare that the family previously received for this child. In addition, child mental health workers will fill out a self-composed questionnaire, with questions about their age, educational background and working experience.

EXPLORATORY MODERATOR VARIABLES

Besides our primary and secondary outcomes (see outcome measures) we will investigate several candidate moderators of treatment effects:

* Parent-reported severity of child disruptive behaviors as measured with the intensity subscale of the Eyberg Child Behavior Inventory (ECBI-I; Robinson et al., 1980);
* Attachment style of parents as measured with the 12-item version of the Revised Experiences in Close Relationship (ECR-R) questionnaire (Wei et al., 2007);
* Parental reward responsivity as measured with the 8-item Reward Responsiveness (RR) questionnaire (Van den Berg et al., 2010);
* Parent-reported child reward responsivity and punishment sensitivity as measured with 22 items of the Sensitivity to Punishment and Sensitivity to Reward Questionnaire for Children (SPSRQ-C) (Luman et al., 2012);
* Parent-reported child differential susceptibility to environmental factors as measured with the 12-item Highly Sensitive Child - Parent Report questionnaire (HSC-PR; Sperati et al., 2022);
* Parent-reported child emotion regulation as measured with the 7-item emotion regulation subscale of the Dutch version of the Behavior Rating Inventory of Executive Function questionnaire (BRIEF-2; Huizinga et al., 2023).

STUDY PROCEDURES

Parents will be recruited within the general practitioners' practices, by child mental health workers or general practitioners. The child mental health worker will inform parents about the study and hand out an information letter. Parents who are interested are asked for verbal consent for the child mental health worker to share their contact information with the researchers. The researchers will use this contact information to further inform parents about the study through telephone calls. If parents want to participate, the researchers will ask them to provide written informed consent. Both legal caretakers (if present) of the child need to provide consent. Parents will have at least 14 days to decide upon participation and ask the researchers any questions. If needed, parents can ask for more time or consult an independent expert to decide upon participation.

After providing informed consent, screening will take place to check whether the family meets all inclusion criteria. If so, parents will be asked to fill in the pre-intervention measurement (T0), whereafter they will be randomized into one of the conditions. A randomization list is generated by and kept by two researchers that are not in any way involved in the study.

To measure the primary and secondary outcomes, parents in both treatment arms will be asked to fill out questionnaires and answer short daily phone calls (at least four days in a row) on a maximum of three measurement occasions. The questionnaires concerning candidate moderators of treatment response will be assessed in both treatment arms during the pre-intervention measurement (T0). The questionnaires will take around 30 minutes to complete at T0, and around 20 minutes at T1 and T2. The daily phone calls will take around two minutes each.

The child mental health workers need to participate in a one-day training provided by two experts in behavioral parent training. Before the one-day training, they are asked to read the materials carefully and to submit a video in which they demonstrate certain aspects of the training. The child mental health workers will receive feedback from the experts or researchers on this video. There are no further requirements that child mental health workers must meet in order to participate, as the group of child mental health workers should be representative for the current situation in general practitioners' practices. Generally, there is a lot of variation between child mental health workers in this setting in terms of study background, years of working experience and postmaster education.

STATISTICAL ANALYSIS

Data will be analyzed on an intention-to-treat basis. Differences in demographic variables between the study-arms will be analyzed with ANOVA's (continuous variables) or chi-squared tests (categorical variables). To examine the effects of the intervention on the primary and secondary outcomes we will conduct multilevel analyses (mixed modeling). Mixed model analysis takes missing data into account (Twisk et al., 2013). We will test a three-level multilevel model: outcomes (level 1), nested within children (level 2) and nested within therapists (level 3). The intercept at therapist level will only be included if the Likelihood Ratio Test shows a significant improvement of the model fit. To assess the influence of exploratory moderating variables on treatment effects, we will include these variables as interaction effects in the multilevel analysis.

ETHICAL CONSIDERATIONS

The risk of any physical or mental harm of the study is very low and not to be expected higher than what may be expected in daily life of the parents and their children. We will exclusively use conventional methods and interventions. The program uses behavioral techniques that were identified as effective for disruptive behaviors in our recent microtrial (Hornstra et al., 2021) and the broader literature (Kaminski et al., 2008; Leijten et al., 2019; Leijten et al., 2021). Parents in both intervention conditions can eventually receive the brief parent training program. Potential adverse reactions will be assessed at T1 (both conditions) and T2 (intervention condition) with a questionnaire. The study is embedded in general practitioners practices.

The children will not be directly involved in the study. They will not be present during the brief parent training sessions and all measures will be parental measures.

Parents can decide to leave the study at any time for any reason if they wish to do so without any consequences.

To debrief participants, parents who wish to learn about the results of the study can request this information from the researchers after the study is finished. This concerns only information on group level. We will inform parents about the possibility to ask for this information in the information letter.

HANDLING AND STORAGE OF DATA AND DOCUMENTS

Digital data, both raw and processed/analyzed data, will be stored at a study specific highly secured folder within the Accare network. This study specific folder can only be accessed by authorized researchers involved in this study.

All questionnaire data, phone call data and audio files (recordings of the sessions) will be stored in one pseudonymized file, that is accompanied by a 'readme' text file that contains a code book explaining the meaning of all variables. The file contains separate pages ("tabs") for all different outcome variables at all different timepoints. A separate logbook-file will be created documenting all decisions that will be made during the process from raw to published data. Old versions of all these documents will be stored, document names will contain their date to ensure version control.

Management of the data and access permissions are with the principal investigator of the research project.

Access permissions are controlled by one of the research project's principal investigators. Raw data containing identifiable information such as the separate log containing participant identification number and study code will be kept strictly separate from the processed data and can only be accessed by the supervisors, research assistants and PhD student. The processed, pseudonymized data will be available for fellow researchers and made available (restricted access) for re-use. Requests for re-use of data after the completion of the research project will be evaluated by principal investigators BvdH, SvdO and TD, who will check whether the research question falls within the scope of the informed consent.

After the research project has been completed (i.e., data collection, data analysis and publishing of research articles completed) all the anonymized (i.e., the link with identifiable information will be deleted) digital data will be transferred to a study specific folder for long-term storage. The folder can only be accessed by the Principal Investigator and by authorized personnel after approval of the principal investigators. This data storage environment allows for careful access management and is only accessible with username and password. Data storage is backed-up automatically daily.

All the research data will be stored for 15 years after the data collection has been completed (i.e. last research assessment for the last participant has been performed). Raw audio-files will be stored for 15 years in an encrypted folder.

TREATMENT INTEGRITY

Intervention integrity will be assessed using procedures based upon work by Abikoff and colleagues (Abikoff et al., 2013; Abikoff et al., 2014). This implies that all intervention sessions will be audiotaped. For every child mental health worker delivering the training, the first session will be checked and child mental health workers will receive feedback on intervention integrity and fidelity by cognitive behavior therapists with extensive experience in behavioral parent training programs. Further, audiotapes of a subset of randomly selected sessions will be scored on intervention integrity and fidelity during the study by independent evaluators. After each session, the child mental health workers have to complete a fidelity checklist in which they will be asked which topics were covered.

ELIGIBILITY:
Inclusion Criteria:

* The child is aged 2 to (until and including) 11 years old;
* Parents have to identify at least four behavioral difficulties of the child at home that they want to target in the training (using the list of 29 target behavioral difficulties (Van den Hoofdakker 2007; Hornstra et al., 2021)).

Exclusion Criteria:

* Current psychotropic medication use of the child (at least not in the month before the training);
* The child has a diagnosis of autism spectrum disorder (as reported by parents, we will not perform any measures to assess autism spectrum disorder);
* The child has an IQ-score of less than 70 (as reported by parents, we will not perform any measures to determine the IQ-score);
* Parents received support or training aimed at remediating behavioral difficulties of the concerned child in the year before the study;
* Not a suitable period for the parents and/or the child to participate in the study (e.g., moving, divorce);
* The child is not living in the same household during at least four weekdays, to ensure that that parent(s) are able to practice the techniques with their child during the week.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Severity of four daily rated target behaviors in specific home situations | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  The primary outcome will be the severity of four parent-rated target behaviors. Parents select four daily occurring behavioral difficulties of the child at home and specific situations in which these behaviors occur. Target behaviors will be selected from an adapted version of a list of 29 possible target behaviors (Hornstra et al., 2021; Van den Hoofdakker et al., 2007), of which parents indicate daily occurrence (yes/no) and (if yes) the severity on a 5-point Likert scale from 1 (not severe) to 5 (extremely severe). Specific situations will be selected from the Home Situation Questionnaire (Breen & Altepeter, 1991). The severity of the four target behaviors within specific situations will be measured with brief daily telephone calls on at least four consecutive school days by the researchers. Parents will be asked whether the four selected target behaviors occurred in the past 24 hours in the selected situation (yes/no) and (if yes) rate the severity on a 5-point Likert scale.

SECONDARY OUTCOMES:
Severity of the same four daily rated target behaviors in other home situations than the specified situation which is used as primary outcome (see primary outcome measure for details on administration) | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  To investigate whether the change in the four target behaviors generalize to other situations, we will also ask parents during the daily phone calls if these behaviors occurred in any of the other situations of the Home Situation Questionnaire (Breen & Altepeter, 1991) in the past 24 hours (yes/no). Items scored as 'yes' will again be rated on a 5-point Likert scale ranging from 1 (not severe) to 5 (extremely severe).
Parent-reported severity of child disruptive behaviors | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  The severity of the child's disruptive behaviors will be assessed with the Intensity subscale of the Eyberg Child Behavior Inventory (ECBI-I; Robinson et al., 1980). The ECBI-I is a questionnaire for parents of children aged 2 to 16, that measures the frequency of 36 child behavior problems on a 7-point Likert scale from 1 (never) to 7 (always).
Parent-reported number of child disruptive behaviors that parents consider as troublesome | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  The number of disruptive behaviors of the child that parents consider as troublesome will be assessed with the Problem subscale of the Eyberg Child Behavior Inventory (ECBI-P; Robinson et al., 1980). The ECBI-P measures whether parents perceive 36 child behavior problems as troublesome on a dichotomous scale with the answer options yes (1) or no (0).
Parent-reported overall impairment of child behavioral difficulties | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  The overall impairment of the child's behavioral difficulties will be assessed with one slightly adapted item of the Impairment Rating Scale (IRS; Fabiano et al., 2006). Parents will be asked to rate the overall severity of their child's behavioral difficulties in functioning and the overall need for treatment, on a 7-point scale ranging from 0 (no problem) to 6 (extreme problem). In the adapted version, we asked parents to specifically link the impairment to the behavioral difficulties.
Parent-reported impact of child behavioral difficulties on the relationship with parents | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  The impact of the child's behavioral difficulties on the relationship with parents will be assessed with one slightly adapted item of the Impairment Rating Scale (IRS; Fabiano et al., 2006). Parents will be asked to rate the impact on a 7-point scale ranging from 0 (no problem) to 6 (extreme problem). In the adapted version, we asked parents to specifically link the impairment to the behavioral difficulties.
Parenting behaviors | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  Parenting behaviors will be assessed with the Alabama Parenting Questionnaire (APQ; Shelton, 1996). The APQ is a 42-item parent-report measure assessing five domains of parenting practices (Involvement, Positive Parenting, Poor Monitoring/Supervision, Inconsistent Discipline, and Corporal Punishment), with 7 additional items (other discipline practices) to prevent negative biases on the domain Corporal Punishment. Parents will rate the items on a 5-point scale ranging from 1 (never) to 5 (always). The APQ total score will be calculated by adding all 35 items from the parenting practices domains. The items from the categories Involvement and Positive Parenting will be recoded. Higher scores therefore indicate less supportive parenting behaviors.
Parenting stress | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  Parenting stress will be assessed with the Parental Stress Scale (PSS; Berry et al., 1995). The PSS is an 18-item parent report scale that measures positive (e.g., emotional benefits) and negative (e.g., restrictions) aspects of parenting. Parents have to agree or disagree with statements concerning parenting on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree).
Parenting self-efficacy and sense of competence | Before randomization (T0), one week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  Parenting self-efficacy will be measured with the Efficacy subscale of the Parenting Sense of Competence Scale (PSOC; Johnston et al., 1989). On the 8 items of this subscale, parents have to rate their capability level and problem-solving ability regarding their parental role on a 6-point Likert scale, ranging from 1 (strongly disagree) to 6 (strongly agree).

OTHER OUTCOMES:
Parents' satisfaction with and opinion about the program | One week after the brief training (experimental arm only) (T1).
  To measure parents' satisfaction with and opinion about the brief parent training, they will be asked to fill in a self-developed satisfaction questionnaire. The questionnaire will be based on questions of the Parent Satisfaction Questionnaire (Bearss et al., 2013), the Therapy Attitude Inventory (Eyberg, 1993; Eyberg & Johnson, 1974), and the questionnaire that was used in Breider and colleagues (2019). Parents have to answer approximately 15 questions about their satisfaction with the brief parent training on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree) and give the brief parent training a grade between 1 (bad) and 10 (good).
Parents' opinions about the acceptability of the program | After the inclusion of participants in the trial is finished, which is anticipated to be in September 2025.
  To measure parents' acceptability about the brief parent training, focus groups will be organized with a number of participating parents. In these groups the new program will be qualitatively evaluated and important information about feasibility, barriers and facilitators for the implementation of the training in general practitioners practices will be gathered.
Child mental health workers' satisfaction with and opinion about the program | After the inclusion of participants in the trial is finished, which is anticipated to be in September 2025.
  To measure child mental health workers' satisfaction with and opinion about the brief parent training, they will be asked to fill in a self-developed satisfaction questionnaire. The questionnaire will be based on questions of the Parent Satisfaction Questionnaire (Bearss et al., 2013), the Therapy Attitude Inventory (Eyberg, 1993; Eyberg & Johnson, 1974), and the questionnaire that was used in Breider and colleagues (2019). Child mental health workers have to answer approximately 15 questions on a 5-point scale ranging from 1 (strongly disagree) to 5 (strongly agree) and give the brief parent training a grade between 1 (bad) and 10 (good).
Child mental health workers' opinions about the acceptability of the program | After the inclusion of participants in the trial is finished, which is anticipated to be in September 2025.
  To measure child mental health workers' acceptability about the brief parent training, focus groups will be organized with a number of therapists, in which important barriers and facilitators for implementation of the program will be identified.
Consumption of other mental healthcare during the trial | One week after the brief training (experimental arm)/eight weeks after T0 (control arm) (T1), three months after T1 (experimental arm only) (T2).
  Potential use of other mental healthcare or support during the trial (T0 to T2) for the behavioral difficulties of the child will be assessed by a self-developed questionnaire, filled out by parents.
Adverse reactions | Three months after T1 (experimental arm only) (T2).
  Potential adverse reactions to the parent training will be measured with a with a self-developed adverse reactions questionnaire filled out by parents. The questionnaire consists of 6 items with the answer options yes or no. If parents answer a question with 'yes' an adverse reaction occurred. In this case, parents will be asked two additional questions for a brief description of the adverse reaction and the time frame.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara J. van den Hoofdakker, Prof. dr., Principal Investigator — Accare Child Study Center; University Medical Center Groningen; University of Groningen; Saskia van der Oord, Prof. dr., Principal Investigator — KU Leuven
Locations (1):
- Accare, Groningen, Netherlands

REFERENCES:
- [Background] Abikoff HB, Thompson M, Laver-Bradbury C, Long N, Forehand RL, Miller Brotman L, Klein RG, Reiss P, Huo L, Sonuga-Barke E. Parent training for preschool ADHD: a randomized controlled trial of specialized and generic programs. J Child Psychol Psychiatry. 2015 Jun;56(6):618-31. doi: 10.1111/jcpp.12346. Epub 2014 Oct 16. PMID 25318650
- [Background] Abikoff H, Gallagher R, Wells KC, Murray DW, Huang L, Lu F, Petkova E. Remediating organizational functioning in children with ADHD: immediate and long-term effects from a randomized controlled trial. J Consult Clin Psychol. 2013 Feb;81(1):113-28. doi: 10.1037/a0029648. Epub 2012 Aug 13. PMID 22889336
- [Background] Bearss K, Johnson C, Handen B, Smith T, Scahill L. A pilot study of parent training in young children with autism spectrum disorders and disruptive behavior. J Autism Dev Disord. 2013 Apr;43(4):829-40. doi: 10.1007/s10803-012-1624-7. PMID 22941342
- [Background] Berry JO, Jones WH. The parental stress scale: Initial psychometric evidence. Journal of Social and Personal Relationships. 1995; 12: 463-472. doi:10.1177/0265407595123009
- [Background] Breen MJ, Altepeter TS. Factor structures of the Home Situations Questionnaire and the School Situations Questionnaire. J Pediatr Psychol. 1991 Feb;16(1):59-67. doi: 10.1093/jpepsy/16.1.59. PMID 2010877
- [Background] Breider S, de Bildt A, Nauta MH, Hoekstra PJ, van den Hoofdakker BJ. Self-directed or therapist-led parent training for children with attention deficit hyperactivity disorder? A randomized controlled non-inferiority pilot trial. Internet Interv. 2019 Aug 8;18:100262. doi: 10.1016/j.invent.2019.100262. eCollection 2019 Dec. PMID 31890615
- [Background] Eyberg S. Consumer satisfaction measures for assessing parent training programs. In VandeCreek L, Knapp S, Jackson TL (Eds.), Innovations in clinical practice: A source book. 1993; 12: 377-382.
- [Background] Eyberg SM, Johnson SM. Multiple assessment of behavior modification with families: effects of contingency contracting and order of treated problems. J Consult Clin Psychol. 1974 Aug;42(4):594-606. doi: 10.1037/h0036723. No abstract available. PMID 4847264
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Fabiano GA, Pelham WE Jr, Waschbusch DA, Gnagy EM, Lahey BB, Chronis AM, Onyango AN, Kipp H, Lopez-Williams A, Burrows-Maclean L. A practical measure of impairment: psychometric properties of the impairment rating scale in samples of children with attention deficit hyperactivity disorder and two school-based samples. J Clin Child Adolesc Psychol. 2006 Sep;35(3):369-85. doi: 10.1207/s15374424jccp3503_3. PMID 16836475
- [Background] Hornstra R, van der Oord S, Staff AI, Hoekstra PJ, Oosterlaan J, van der Veen-Mulders L, Luman M, van den Hoofdakker BJ. Which Techniques Work in Behavioral Parent Training for Children with ADHD? A Randomized Controlled Microtrial. J Clin Child Adolesc Psychol. 2021 Nov-Dec;50(6):888-903. doi: 10.1080/15374416.2021.1955368. Epub 2021 Aug 23. PMID 34424102
- [Background] Huizinga M, Smidts DP. Age-related changes in executive function: A normative study with the Dutch version of the Behavior Rating Inventory of Executive Function (BRIEF). Child Neuropsychol. 2011;17(1):51-66. doi: 10.1080/09297049.2010.509715. PMID 21218296
- [Background] Johnston C, Mash EJ. A Measure of Parenting Satisfaction and Efficacy. Journal of Clinical Child Psychology. 1989; 18(2): 167-175. doi:10.1207/s15374424jccp1802_8
- [Background] Kaminski JW, Claussen AH. Evidence Base Update for Psychosocial Treatments for Disruptive Behaviors in Children. J Clin Child Adolesc Psychol. 2017 Jul-Aug;46(4):477-499. doi: 10.1080/15374416.2017.1310044. Epub 2017 May 1. PMID 28459280
- [Background] Kaminski JW, Valle LA, Filene JH, Boyle CL. A meta-analytic review of components associated with parent training program effectiveness. J Abnorm Child Psychol. 2008 May;36(4):567-89. doi: 10.1007/s10802-007-9201-9. Epub 2008 Jan 19. PMID 18205039
- [Background] Leijten P, Gardner F, Melendez-Torres GJ, van Aar J, Hutchings J, Schulz S, Knerr W, Overbeek G. Meta-Analyses: Key Parenting Program Components for Disruptive Child Behavior. J Am Acad Child Adolesc Psychiatry. 2019 Feb;58(2):180-190. doi: 10.1016/j.jaac.2018.07.900. Epub 2018 Nov 26. PMID 30738545
- [Background] Leijten P, Melendez-Torres GJ, Gardner F. Research Review: The most effective parenting program content for disruptive child behavior - a network meta-analysis. J Child Psychol Psychiatry. 2022 Feb;63(2):132-142. doi: 10.1111/jcpp.13483. Epub 2021 Jul 9. PMID 34240409
- [Background] Luman M, van Meel CS, Oosterlaan J, Geurts HM. Reward and punishment sensitivity in children with ADHD: validating the Sensitivity to Punishment and Sensitivity to Reward Questionnaire for children (SPSRQ-C). J Abnorm Child Psychol. 2012 Jan;40(1):145-57. doi: 10.1007/s10802-011-9547-x. PMID 21789519
- [Background] Robinson EA, Eyberg SM, Ross AW. The standardization of an inventory of child conduct problem behaviors. Journal of Clinical Child & Adolescent Psychology. 1980; 9(1): 22-28. doi:10.1080/15374418009532938
- [Background] Shelton KK, Frick PJ, Wootton J. Assessment of Parenting Practices in Families of Elementary School-Age Children. Journal of Clinical Child Psychology. 1996; 25: 317-329. doi:10.1207/s15374424jccp2503_8
- [Background] Sperati A, Spinelli M, Fasolo M, Pastore M, Pluess M, Lionetti F. Investigating sensitivity through the lens of parents: validation of the parent-report version of the Highly Sensitive Child scale. Dev Psychopathol. 2024 Feb;36(1):415-428. doi: 10.1017/S0954579422001298. Epub 2022 Dec 12. PMID 36503569
- [Background] Twisk J, de Boer M, de Vente W, Heymans M. Multiple imputation of missing values was not necessary before performing a longitudinal mixed-model analysis. J Clin Epidemiol. 2013 Sep;66(9):1022-8. doi: 10.1016/j.jclinepi.2013.03.017. Epub 2013 Jun 21. PMID 23790725
- [Background] Van den Berg I, Franken IH, Muris P. A new scale for measuring reward responsiveness. Front Psychol. 2010 Dec 31;1:239. doi: 10.3389/fpsyg.2010.00239. eCollection 2010. PMID 21922010
- [Background] van den Hoofdakker BJ, van der Veen-Mulders L, Sytema S, Emmelkamp PMG, Minderaa RB, Nauta MH. Effectiveness of behavioral parent training for children with ADHD in routine clinical practice: a randomized controlled study. J Am Acad Child Adolesc Psychiatry. 2007 Oct;46(10):1263-1271. doi: 10.1097/chi.0b013e3181354bc2. PMID 17885567
- [Background] Wei M, Russell DW, Mallinckrodt B, Vogel DL. The Experiences in Close Relationship Scale (ECR)-short form: reliability, validity, and factor structure. J Pers Assess. 2007 Apr;88(2):187-204. doi: 10.1080/00223890701268041. PMID 17437384